CLINICAL TRIAL: NCT02362347
Title: Investigating Novel Treatments for Concussion: Impact of Compression Vest on Rehabilitation Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western University, Canada (Other)
Collaborators: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Kevin Shoemaker, Professor, PhD, Western University, Canada
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CON001
Record Dates: First submitted 2015-02-05; First posted 2015-02-12 (Estimated); Last update posted 2019-03-06 (Actual); Status verified 2019-03

CONDITIONS: Brain Concussion; Post-Concussion Syndrome
MeSH Terms: conditions — Brain Concussion; Post-Concussion Syndrome | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Usual care + exercise (Active Comparator): Usual care + exercise
  Interventions: Other: exercise
- No care, no exercise (No Intervention): No care, no exercise
- Usual care + exercise + compression vest (Experimental): Usual care + exercise + London Health Sciences Centre - Compression Vest
  Interventions: Device: London Health Sciences Centre - Compression Vest; Other: exercise

INTERVENTIONS:
Device: London Health Sciences Centre - Compression Vest — London Health Sciences Centre - Compression Vest
  Arms: Usual care + exercise + compression vest
Other: exercise — exercise
  Arms: Usual care + exercise; Usual care + exercise + compression vest

SUMMARY:
The purpose of this investigation is to determine the effect of a weighted compression vest in addition to usual medical care and exercise rehabilitation on cardiovascular, neurocognitive, balance and anxiety measures in individuals medically diagnosed with, and being treated for, a mild traumatic brain injury.

DETAILED DESCRIPTION:
Mild traumatic brain injury (mTBI), or concussion, induces significant impairment to a patient's mobility and tolerance for daily living activities with symptoms that include decreased balance, dizziness, confusion, headaches, visual and auditory sensitivities. If recognized promptly, many of these injuries respond well to immediate rest and standard rehabilitation strategies. However, approximately 10-30% of these patients will experience persistent symptoms beyond the ~2 week period of spontaneous healing. The persistent symptoms point to neural damage, or disrupted neural networks in the brain, but the actual mechanism or nature of neural damage remains to be elucidated. The brain's neural activity must be supported by rapid adjustments to, and optimal distribution of, blood flow. However, cerebrovascular control remains poorly studied in the context of persistent concussion symptoms, particularly the reactivity element of flow control such as how fast it recovers during drops in blood pressure such as when one stands up from the sitting posture. Cerebrovascular damage in mTBI appears to affect mostly the autoregulatory adjustments to changes in brain perfusion pressure (i.e., from lying down to standing up) (Len et al., 2013;Junger et al., 1997). The investigators will study the impact of mTBI in both acute and persistent stages on cerebrovascular adjustments to metabolic and pressure-dependent stimuli. Currently, decisions regarding rate and completeness of healing remain subjective which can lead to earlier-than-optimal return of the patient to inappropriate levels of activity, work or school. Improved and cost-effective markers of the rate and completeness of brain healing are needed that can be obtained in the clinic. One challenge might be the emphasis in previous investigations on searching for a single biomarker of damage in a highly integrated system. Rather, the investigators believe it may be more effective to employ a holistic perspective; focusing on a comprehensive neural outcome might provide enhanced insight into the severity of damage and rate or completion of recovery. Previously, several investigators established heart rate variability (HRV) as sensitive marker of abnormal brain function in TBI (traumatic brain injury) cases for both adults and children (Goldstein et al., 1998;Goldstein et al., 1996). Moreover, these studies imply that autonomic nervous system control of heart rate is disrupted in proportion to the degree of neurologic insult. Thus, heart rate power spectral analysis may prove to be a useful adjunct in determining severity of neurologic injury and prognosis for recovery. Despite many studies outlining the relationship between mTBI and HRV (Ryan et al., 2011;Goldstein et al., 1998;Goldstein et al., 1996;Papaioannou et al., 2008;La Fountaine et al., 2009) no follow-up research has been conducted to establish this method (which is cost-effective, non-invasive, comprehensive and easily-obtained) as a routine assessment of TBI severity, or rehabilitative efficacy. An additional neural network associated with cardiac function is the baroreflex and the sensitivity of this neural network (baroreflex sensitivity; BRS) can be studied with non-invasive measures of heart rate and blood pressure. In the past and currently our lab has used both methods of HRV and BRS safely and effectively (Zamir et al., 2013;Kiviniemi et al., 2010;Kiviniemi et al., 2011;Shoemaker et al., 2012). This current study will assess the feasibility and impact of routine measurements of cardiac dynamics as a sensitive marker of the severity and persistence of "overall" brain damage in mTBI patients. Based on more than 30 failed clinical trials, no single pharmacological agent can be prescribed to minimize TBI-induced brain damage, despite efficacy shown for several agents in rodent studies (see (Kabadi & Faden, 2014) for review). In contrast, non-pharmacological approaches in rodents, show that both pathophysiological changes and neurological impairment after experimental TBI can be attenuated by physical activity (Griesbach et al., 2004;Griesbach et al., 2009). Thus, there is value in considering application of "appropriate" exercise as soon as possible in mTBI patients, but not too soon because the value of exercise in rodent models were observed only when applied after the acute stage (Griesbach et al., 2007;Piao et al., 2013). Therefore, this study will also examine the impact of adding prescriptive exercise in addition to usual clinical care on the rate of concussion recovery. Enabling patients to receive the benefits of enhanced levels of physical activity during treatments for concussion may be limited by the concussion symptoms. Nonetheless, recent anecdotal evidence from our Parkwood group has illustrated the remarkable benefit to many patients with persistent symptoms provided by the wearing of a compression vest (HSREB #103325 and #104865). Briefly, the weighted compression vests (5% of the individual's body mass) are individualized and fitted to each subject to ensure its snug but does not impede one's respirations (similar to a bulletproof vest). The noted benefits of the compression vest include instant improvements to balance and gait, and reduced anxiety during stair climbing. Since this adaptive method of treatment appears to exert a powerful effect on enhancing patient's ability to perform exercise, and is consistent with the personalized medicine approach (like the exercise intervention), further investigation into the effect of the compression vest on concussion symptoms and rehabilitation is a viable area of research. To date the impact of compression vest interventions has yet to be examined in patients during the acute TBI phase or in younger individuals. Thus, the aim of the next phase of study is to establish whether interventions with a weighted compression vest can enhance exercise tolerance for patients in both acute and persistent phases of the TBI, with explorations into possible mechanistic links to cerebrovascular, cardiovascular and neural outcomes. If so, then new evidence supporting the use of compression vests could change clinical practice and, importantly, improve long-term health outcomes for many patients. In review, the purpose of this investigation is to determine the efficacy of novel methods of mild traumatic brain injury rehabilitation in addition to usual concussion rehabilitation programs. Concussed participants will complete a longitudinal study in which they will be randomly allocated to one of three rehabilitation groups: 1) usual care 2) usual care + exercise 3) usual care + exercise + compression vest. The efficacy of each rehabilitation group will be primarily quantified via changes in routine cardiac dynamic measurements (HRV, BRS, changes in blood flow with changes in posture).

ELIGIBILITY:
Inclusion Criteria:

* concussed: medically diagnosed with, and being treated for a concussion for no longer than 1 year
* healthy volunteer: no previous medical diagnosis of a concussion

Exclusion Criteria:

* bone or muscle problems that could impact balance or how well you walk
* diagnosis of pre-existing heart disease
* medications that affect heart or blood vessel control
* pre-existing brain disorders such as Parkinson's, Multiple Sclerosis, Raynaud's, Multiple System Atrophy, metabolic disorders such as diabetes, a history of significant neck injury, or focal neurologic deficit
* primary or metastatic bone tumour
* severe osteoporosis
* if you are, or think you might be, pregnant or breastfeeding
* if you are not able to be understand English

Ages: 12 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 153 (Actual)
Dates: Start 2015-02; Primary Completion 2019-03-04 (Actual); Study Completion 2019-03-04 (Actual)

PRIMARY OUTCOMES:
Change in symptom profile | baseline, two-weeks, three-weeks, four-weeks, 5-weeks and 6-weeks post-baseline
  Timeline to asymptomatic and clinical discharge
Change in exercise tolerance | baseline, four-weeks post-baseline, six-week post-baseline
  Duration and wattage achieved at symptom exacerbation

SECONDARY OUTCOMES:
Anxiety | baseline, two-weeks, three-weeks, four-weeks, 5-weeks and 6-weeks post-baseline
  Generalized Anxiety Disorder 7-item (GAD-7) scale
Balance | baseline, two-weeks, three-weeks, four-weeks, 5-weeks and 6-weeks post-baseline
  Change in Stability Index, quantified via BioDex Technology
Transcranial Doppler Ultrasound - Cerebrovascular Function | baseline, two-weeks, three-weeks, four-weeks, 5-weeks and 6-weeks post-baseline
  Change in middle cerebral artery blood velocity - cm/s
Heart Rate Variability | baseline, two-weeks, three-weeks, four-weeks, 5-weeks and 6-weeks post-baseline
  Measure of autonomic function - quantified via R-R interval duration (seconds)
Baroreflex Sensitivity | baseline, two-weeks, three-weeks, four-weeks, 5-weeks and 6-weeks post-baseline
  Measure of autonomic function - quantified via changes in blood pressure for a given heart rate
Cognitive Function | baseline, two-weeks, three-weeks, four-weeks, 5-weeks and 6-weeks post-baseline
  Cogingram - assessment of psychomotor function, attention, learning and working memory

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Shoemaker, PhD, Principal Investigator — Western University
Locations (2):
- Canada (2):
  - Fowler Kennedy Sports Medicine Clinic, London, Ontario
  - Neurovascular Research Laboratory, London, Ontario

REFERENCES:
- [Background] Goldstein B, Kempski MH, DeKing D, Cox C, DeLong DJ, Kelly MM, Woolf PD. Autonomic control of heart rate after brain injury in children. Crit Care Med. 1996 Feb;24(2):234-40. doi: 10.1097/00003246-199602000-00009. PMID 8605794
- [Background] Goldstein B, Toweill D, Lai S, Sonnenthal K, Kimberly B. Uncoupling of the autonomic and cardiovascular systems in acute brain injury. Am J Physiol. 1998 Oct;275(4):R1287-92. doi: 10.1152/ajpregu.1998.275.4.R1287. PMID 9756562
- [Background] Griesbach GS, Gomez-Pinilla F, Hovda DA. Time window for voluntary exercise-induced increases in hippocampal neuroplasticity molecules after traumatic brain injury is severity dependent. J Neurotrauma. 2007 Jul;24(7):1161-71. doi: 10.1089/neu.2006.0255. PMID 17610355
- [Background] Griesbach GS, Hovda DA, Gomez-Pinilla F. Exercise-induced improvement in cognitive performance after traumatic brain injury in rats is dependent on BDNF activation. Brain Res. 2009 Sep 8;1288:105-15. doi: 10.1016/j.brainres.2009.06.045. Epub 2009 Jun 23. PMID 19555673
- [Background] Griesbach GS, Hovda DA, Molteni R, Wu A, Gomez-Pinilla F. Voluntary exercise following traumatic brain injury: brain-derived neurotrophic factor upregulation and recovery of function. Neuroscience. 2004;125(1):129-39. doi: 10.1016/j.neuroscience.2004.01.030. PMID 15051152
- [Background] Junger EC, Newell DW, Grant GA, Avellino AM, Ghatan S, Douville CM, Lam AM, Aaslid R, Winn HR. Cerebral autoregulation following minor head injury. J Neurosurg. 1997 Mar;86(3):425-32. doi: 10.3171/jns.1997.86.3.0425. PMID 9046298
- [Background] Kabadi SV, Faden AI. Neuroprotective strategies for traumatic brain injury: improving clinical translation. Int J Mol Sci. 2014 Jan 17;15(1):1216-36. doi: 10.3390/ijms15011216. PMID 24445258
- [Background] Kiviniemi AM, Frances MF, Tiinanen S, Craen R, Rachinsky M, Petrella RJ, Seppanen T, Huikuri HV, Tulppo MP, Shoemaker JK. alpha-Adrenergic effects on low-frequency oscillations in blood pressure and R-R intervals during sympathetic activation. Exp Physiol. 2011 Aug;96(8):718-35. doi: 10.1113/expphysiol.2011.058768. Epub 2011 May 20. PMID 21602293
- [Background] Kiviniemi AM, Tiinanen S, Hautala AJ, Seppanen T, Makikallio TH, Huikuri HV, Tulppo MP. Frequency of slow oscillations in arterial pressure and R-R intervals during muscle metaboreflex activation. Auton Neurosci. 2010 Jan 15;152(1-2):88-95. doi: 10.1016/j.autneu.2009.08.020. Epub 2009 Sep 19. PMID 19767247
- [Background] La Fountaine MF, Heffernan KS, Gossett JD, Bauman WA, De Meersman RE. Transient suppression of heart rate complexity in concussed athletes. Auton Neurosci. 2009 Jun 15;148(1-2):101-3. doi: 10.1016/j.autneu.2009.03.001. Epub 2009 Mar 21. PMID 19303821
- [Background] Len TK, Neary JP, Asmundson GJ, Candow DG, Goodman DG, Bjornson B, Bhambhani YN. Serial monitoring of CO2 reactivity following sport concussion using hypocapnia and hypercapnia. Brain Inj. 2013;27(3):346-53. doi: 10.3109/02699052.2012.743185. PMID 23438354
- [Background] Papaioannou V, Giannakou M, Maglaveras N, Sofianos E, Giala M. Investigation of heart rate and blood pressure variability, baroreflex sensitivity, and approximate entropy in acute brain injury patients. J Crit Care. 2008 Sep;23(3):380-6. doi: 10.1016/j.jcrc.2007.04.006. Epub 2007 Dec 11. PMID 18725044
- [Background] Piao CS, Stoica BA, Wu J, Sabirzhanov B, Zhao Z, Cabatbat R, Loane DJ, Faden AI. Late exercise reduces neuroinflammation and cognitive dysfunction after traumatic brain injury. Neurobiol Dis. 2013 Jun;54:252-63. doi: 10.1016/j.nbd.2012.12.017. Epub 2013 Jan 8. PMID 23313314
- [Background] Ryan ML, Ogilvie MP, Pereira BM, Gomez-Rodriguez JC, Manning RJ, Vargas PA, Duncan RC, Proctor KG. Heart rate variability is an independent predictor of morbidity and mortality in hemodynamically stable trauma patients. J Trauma. 2011 Jun;70(6):1371-80. doi: 10.1097/TA.0b013e31821858e6. PMID 21817974
- [Background] Shoemaker JK, Usselman CW, Rothwell A, Wong SW. Altered cortical activation patterns associated with baroreflex unloading following 24 h of physical deconditioning. Exp Physiol. 2012 Dec;97(12):1249-62. doi: 10.1113/expphysiol.2012.065557. Epub 2012 May 21. PMID 22613740